CLINICAL TRIAL: NCT04693104
Title: Effects of PVA Hydrogel in Comparison With Synvisc-One®, in Patients With Knee Osteoarthritis
Brief Title: Intra-articular PVA Hydrogel in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rottapharm Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PVA-001
Record Dates: First submitted 2020-12-27; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Given the impossibility of obtaining identical presentations of the compared interventions, double-blind conditions will be ensured by appointing at each site one "injector investigator" in charge only of the administration of the treatments and one "clinical assessor investigator" as Outcome Assessor, in charge of all safety and efficacy assessments, who will remain always blinded to the treatment. Patient blinding will be ensured by avoiding visual access to the injection field by the use of a screen between the patient and his/her knee.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVA Hydrogel (Experimental): PVA Hydrogel (Rottapharm Biotech, Monza): 2 mL prefilled syringe for intra-articular injection
  Interventions: Device: PVA Hydrogel
- Synvisc-One® (Active Comparator): Synvisc-One® (Genzyme Corporation, Ridegield, New Jersey, USA): 6 mL prefilled syringe for intra-articular injection
  Interventions: Device: Synvisk-One®

INTERVENTIONS:
Device: PVA Hydrogel — PVA Hydrogel will be supplied in 2 mL sterile and endotoxins-free pre-filled syringes containing a biocompatible polyvinyl alcohol crosslinked (PVA CL, main component) and buffered water for injections.
  Arms: PVA Hydrogel
Device: Synvisk-One® — Synvisc One® (comparator) will be supplied in a 6 mL sterile and non-pyrogenic syringe containing containing Hylan polymers (hylan A + hylan B) (main component), sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate monohydrate and water for injections.
  Arms: Synvisc-One®

SUMMARY:
This multicentre, prospective, randomized, double-blind, active-controlled, parallel group clinical investigation is aimed to assess the safety and the clinical performance over 6 months of a single intra-articular injection of PVA Hydrogel, novel polyvinyl alcohol preparation, as compared to hyalan G-F20, (Synvisc-One®) one of the most commonly used and best performing hyaluronic acid based products, in patients with symptomatic knee osteoarthitis (OA).

DETAILED DESCRIPTION:
To compare the effects of a single intra-articular injection of a novel polyvinyl alcohol preparation (PVA Hydrogel) and hylan G-F20 (Synvisc-One®) in patients with symptomatic knee OA.

Patients with knee OA (ACR clinical and radiological criteria) symptoms for ≥6 months, insufficient/failed response to analgesics, K&L stage II-III (x-Rays within past 12 months), a knee pain score of 4-9 (0-10 NRS) in the target knee and <3 in the contralateral knee, will be enrolled in a randomised, controlled, double-blind, parallel group 26-week clinical investigation to receive a single intra-articular injection of PVA Hydrogel or Synvisc-One®. Safety (both at the injection site (primary end-point) and overall) and efficacy (change in pain in the target knee (0-10 NRS), WOMAC Osteoarthritis Index (total and subscales) and Patient's Global Assessment of knee OA (0-10 NRS)) will be evaluated.

After signing an informed consent, patients will be screened at least 7 days before randomisation, when they will received a single intra-articular injection of either PVA Hydrogel or Synvisc-One® (1:1 allocation ratio) and will be then seen for follow-up 1, 2 and 4 days (this latter just in case of AE occurrence at the target knee) and 2, 4, 8, 12, 18 and 26 weeks after IA injection.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before undergoing any clinical-investigation-related procedure.
2. Male or female aged between 40 and 80 years.
3. Documented diagnosis of primary OA of the knee, based on the clinical and radiological American College of Rheumatology (ACR) criteria for knee OA:

   * Knee pain,
   * X-ray osteophytes,
   * at least one of the following: (a) age >50 years; (b) morning stiffness <30 minutes in duration; (c) crepitus on active motion.
4. Grade II-III according to the Kellgren and Lawrence classification (X-ray evidence at enrolment or within the previous 12 months).
5. Knee OA symptoms for at least six months.
6. Failure to respond (i.e. did not respond sufficiently) to analgesics and/or regular NSAIDs, or proven intolerance to regular use of NSAIDs or to weak opioids analgesics.
7. Presence of pain in the target knee, with a value ≥4 and ≤9 on the NRS, providing that pain in the contralateral knee I less than 3 (see also Exclusion Criteria n. 3).
8. Ability and willingness to communicate, participate, and comply with the requirements and scheduled procedures of the clinical investigation.

Exclusion Criteria:

(a) Medical history and Concomitant Diseases related criteria

1. Presence of isolated or predominantly symptomatic patellofemoral OA of the knee (i.e. pain when climbing stairs or forcing the patient to extend his leg when sitting on a low sit).
2. Presence of secondary osteoarthritis and/or other rheumatic diseases. In particular, history or presence of the following diseases should be excluded: septic arthritis, inflammatory joint disease, gout, recurrent episodes of pseudogout, Paget's disease of bone, articular fracture, ochronosis, acromegaly, haemocromatosis, Wilson's disease, primary osteochondromatosis.
3. Contralateral (i.e. non-target) knee pain >3 on the NRS
4. Any knee OA treatment for both knees (other than the clinical investigation viscosupplementation of the target knee) anticipated within the next 6 months.
5. Presence of pain (any severity) in the ipsilateral and/or contralateral hip.
6. Presence of disease of the spine or other lower extremity joints of sufficient severity to affect the clinical investigation assessments.
7. Anterior cruciate ligament repair, reconstruction or injury in the target knee within the previous 3 years.
8. Cartilage repair/surgery in the target knee within the previous 3 years.
9. Any surgery in the lower limbs within the previous 12 months
10. Any planned surgery of the lower limbs during the clinical investigation period.
11. Significant articular deformities of the lower limbs, i.e. major dysplasia and congenital abnormalities.
12. Presence of varus or valgus knee deformity ≥ 8°.
13. History or presence of osteonecrosis in the lower limbs.
14. Presence of any significant injury of the ipsilateral limb within the previous 6 months.
15. Presence of joint effusion and/or infection at the target knee.
16. Presence of local skin abnormalities (e.g. infection or disease) at the target knee.
17. History or presence of knee joint infection secondary to previous intra-articular injections, or increased predisposition to infections.
18. History or high risk of venous thromboembolism and/or venous or lymphatic stasis of the limb of the target knee.
19. History of allergy or known hypersensitivity to hyaluronic acid, to any of the components of the products under clinical investigation, or to paracetamol.
20. History of hypersensitivity to avian proteins.
21. Morbidly obese patients (BMI≥35).
22. Severe concomitant disease at any organ or apparatus (including acute or chronic infectious diseases) that may interfere with the free use and evaluation of the affected knee for the 6 months course of the clinical investigation and/or malignancy (with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin or in situ uterine cervical cancer) active within the previous 12 months.
23. History of drug, alcohol, or other substance abuse, or other factors limiting the ability to cooperate during the clinical investigation.
24. Any other clinically relevant disease and condition that, in the opinion of the principal investigators, may jeopardize the clinical investigation conduct according to the CIP or performance or safety assessments or may compromise the patients' safety or may place the patient at an undue risk by participating in the clinical investigation.

    (b) Previous or concomitant treatments
25. Patients requiring systemic analgesics (including opiates)/NSAIDs for the target knee, or for indications other than OA pain at the target knee but likely to use these medications for more than 5 consecutive days, or for more than 10 non-consecutive days in one month, or unable to stop them during the 2 days preceding a clinic visit.
26. Patients requiring topical analgesics/NSAIDs for the target knee.
27. Patient requiring intra-articular corticosteroids into any joint or periarticular structure in the lower limb, or systemic corticosteroids (oral or injected for any indication).
28. Patients who underwent tidal lavage of the knee joint(s) during the three months prior to randomization.
29. Viscosupplementation in the lower limbs within the previous 12 months.
30. Patients on SYSADOAs or a dietary supplement containing compounds considered specific for OA (e.g. glucosamine, chondroitin sulphate, diacerein) if the dosage has not been stable within the previous 3 months.
31. Patients on anticoagulant treatment other than direct oral anticoagulants (DOACS).
32. Non-pharmacological therapy for the lower extremities, unless stable for more than one month (and not to be substantially altered during the clinical investigation). Physical therapy is allowed.
33. Patients using assistive devices other than a cane (walking stick) or knee brace.
34. Concomitant participation in any clinical study/investigation or treatment with any investigational drugs/treatments/devices within the previous 3 months or 5 of half-lives (whichever is longer).
35. Contraindication to use of hyaluronic acid.
36. Contraindication to use of paracetamol. (c) Other
37. For women of childbearing potential, not surgically sterile or postmenopausal:

    * Pregnancy (i.e. positive pregnancy test at screening) or breastfeeding;
    * Failure to agree to practice a highly effective method of contraception for 3 months after the IA injection.
38. For sexually active men with a female partner of childbearing potential: failure to use a reliable method of birth control for 3 months after the IA injection.

Randomization Criteria:

1. Pain value in the target knee ≥4 and ≤9 on the NRS.
2. Absence of joint effusion in the target knee.
3. Absence of local skin abnormalities (e.g. infection or disease) at the target knee.
4. No use of analgesics/NSAIDs during the 2 days preceding the Randomization Visit.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Adverse Events at the injection site (target knee) | 6 months
  patient reported symptom and/or investigator detected clinical sign
Adverse Device Events | 6 months
  AEs considered as related to the device and/or to the IA procedure.

SECONDARY OUTCOMES:
Device Deficiencies | 6 months
  malfunctions, use errors and inadequate labelling occurred before, during or after the use of the devices
Adverse Events | 6 months
  any AE irrespective of target knee involvement
Physical examination | 6 months
  a complete physical examination will be carried out at all scheduled clinic visits and/or at any unscheduled/early termination visit in case of premature discontinuation. Clinically significant findings of the physical examination at screening will be documented as concomitant diseases. New findings or worsening of a finding at all visits following the screening visit will recorded as adverse events.
Blood pressure | 6 months
  Systolic and diastolic blood pressure (mmHg)
Pulse rate | 6 months
  Radial pulse rate (beats/minute)
Body temperature | 6 months
  Body temperature will be assessed via a mouth thermometer (degrees Celsius (°C)
Knee pain | 6 months
  0-10 NRS ("0=no pain" to "10=the worst possible pain") during past 48 hours
WOMAC Index | 6 months
  tri-dimensional, disease-specific, self-administered, health status measure, to assess pain, stiffness and physical function in patients with knee OA, NRS format, version 3.1, 48 hours recall period
Patient's Global Assessment of knee OA | 6 months
  overall judgment of efficacy ("Considering all the ways your knee osteoarthritis affects you, how would you rate the severity of your condition over the last week?" according to a 0-10 NRS scale, anchored at 0 = "I am feeling very well" and 10 = "I am feeling as bad as possible"
Rescue medication use | 6 months
  Number of paracetamol tablets taken each day

CONTACTS AND LOCATIONS:
Overall Officials: Tomaz Blicharski, Study Director — Lubelskie Centrum Diagnostyczne, Swidnik, Poland
Locations (1):
- Lubelskie Centrum Diagnostyczne, Świdnik, Poland

IPD SHARING:
Plan to Share IPD: No